CLINICAL TRIAL: NCT01616082
Title: Effect of Caloric Restriction on Metabolic Biomarkers and Fat Oxidation in Obese Men and Women (Magellan II)
Brief Title: Effect of Caloric Restriction on Fat Oxidation in Obese Men and Women (Magellan II)
Acronym: MagellanII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMDFH 266040; 266040 (Other: Florida Hospital IRB)
Record Dates: First submitted 2012-06-04; First posted 2012-06-11 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Obesity; Overweight; Metabolic Diseases
Keywords: fatty acid oxidation; Proton magnetic resonance spectroscopy
MeSH Terms: conditions — Obesity; Overweight; Metabolic Diseases | interventions — Caloric Restriction; Phentermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Overwight/Obese with no drug (Active Comparator): After screening, overweight/obese subjects (BMI >27 - ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved.
  Interventions: Behavioral: Low Calorie Diet (LCD)
- Overweight/obese with Phentermine (Active Comparator): After screening, overweight/obese (BMI >27.0 - ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved. Individuals not on track to achieve their target weight by four weeks will receive the drug Phentermine to promote weight loss. Then, following eight weeks LCD (or four weeks LCD + four weeks LCD+Phentermine), in the event that they did not achieve the target weight loss, subjects will be given the option to continue with the LCD + Phentermine for up to an additional 12 weeks, under a doctor's supervision.
  Interventions: Behavioral: Low Calorie Diet (LCD); Drug: Phentermine

INTERVENTIONS:
Behavioral: Low Calorie Diet (LCD) — A Diet History Questionnaire was completed and subjects had dietary counseling and were provided shakes. The low calorie diet began, to continued for a period of 8 weeks.
Drug: Phentermine — Individuals not on track to achieve their target weight by four weeks received the drug Phentermine to promote weight loss. Then, following eight weeks LCD (or four weeks LCD + four weeks LCD+Phentermine), in the event that they did not achieve the target weight loss, subjects were given the option to continue with the LCD + Phentermine for up to an additional 12 weeks, under a doctor's supervision.
  Protection Against Risk:
  * Prior to administering any phentermine, a history and physical including EKG will be conducted (at the screening visit) and will be used to determine whether the participant is clear to receive the medication.
  * Participants will see the study doctor or nurse practitioner at every study visit after the drug is initiated.
  Arms: Overweight/obese with Phentermine

SUMMARY:
The purpose of this study is to better understand the different ways our bodies burn fat which may be important for obesity, diabetes, and cardiovascular disease.

DETAILED DESCRIPTION:
In this study the investigators will examine the hypothesis that overweight/obese individuals that are unable to meet target weight loss goals on a low calorie diet (LCD) are intrinsically less metabolically flexible than their weight-losing counterparts. The investigators expect that this 'inflexibility' will be characterized by impaired fat oxidation (as determined by indirect calorimetry) in response to caloric restriction. If this were the case, these subjects may represent a population of 'super-responders' likely to demonstrate a robust response to approaches to increase fat oxidation. The investigators will also measure lipid concentrations in skeletal muscle and liver by hydrogen 1 magnetic resonance (1H-MRS) to determine both the stability of these measurements as well as the magnitude of changes that can be seen during LCD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) 27-30 kg/m2, inclusive, with hypertension, controlled (<140 / <90) either by diet or medication.
* BMI 30-40 kg/m2, inclusive.
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (hypertension controlled (<140 / <90) either by diet or medication is acceptable), hepatic, psychiatric, neurologic, allergic, (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing), muscle disease, diabetes, or severe uncontrolled hypertension.
* Known hypersensitivity to phentermine, lidocaine, bupivicaine or any medication component of the study procedure.
* Presence of cardiac pacemaker, implanted cardiac defibrillator, or brain aneurysm clips.
* Any significant bleeding diathesis which could preclude recovery from the biopsy procedure. ASA, ibuprofen, and any other oral anti platelet agent will be discontinued at least 7 days prior to procedure.
* Abnormal CK as per site laboratory ranges.
* Subjects with either a medical history of or physical evidence of keloid scar formation upon physical examination.
* 12-lead electrocardiogram (ECG) demonstrating a clinically significant abnormality.
* Pregnant or nursing females or females less than 6 months postpartum from the scheduled date of collection.
* Participation in non-routine rigorous exercise (e.g., road races, heavy lifting, etc.) within one week prior to the muscle biopsy procedures.
* Presence of any condition in the investigator's opinion that may negatively affect subject safety or protocol adherence.
* Females of childbearing potential (any female except those with tubal ligation, hysterectomy, or absence of menses > 2years) unwilling to use an approved method of contraception (condom, diaphragm, implantable uterine device (IUD) that does not release hormones).
* Prior participation in the Magellan I study at the Translational Research Institute for Metabolism and Diabetes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Holloway GP, Bonen A, Spriet LL. Regulation of skeletal muscle mitochondrial fatty acid metabolism in lean and obese individuals. Am J Clin Nutr. 2009 Jan;89(1):455S-62S. doi: 10.3945/ajcn.2008.26717B. Epub 2008 Dec 3. PMID 19056573
- [Background] Simoneau JA, Kelley DE. Altered glycolytic and oxidative capacities of skeletal muscle contribute to insulin resistance in NIDDM. J Appl Physiol (1985). 1997 Jul;83(1):166-71. doi: 10.1152/jappl.1997.83.1.166. PMID 9216960
- [Background] Ukropcova B, Sereda O, de Jonge L, Bogacka I, Nguyen T, Xie H, Bray GA, Smith SR. Family history of diabetes links impaired substrate switching and reduced mitochondrial content in skeletal muscle. Diabetes. 2007 Mar;56(3):720-7. doi: 10.2337/db06-0521. PMID 17327442
- [Background] Zurlo F, Lillioja S, Esposito-Del Puente A, Nyomba BL, Raz I, Saad MF, Swinburn BA, Knowler WC, Bogardus C, Ravussin E. Low ratio of fat to carbohydrate oxidation as predictor of weight gain: study of 24-h RQ. Am J Physiol. 1990 Nov;259(5 Pt 1):E650-7. doi: 10.1152/ajpendo.1990.259.5.E650. PMID 2240203
- [Background] Koves TR, Ussher JR, Noland RC, Slentz D, Mosedale M, Ilkayeva O, Bain J, Stevens R, Dyck JR, Newgard CB, Lopaschuk GD, Muoio DM. Mitochondrial overload and incomplete fatty acid oxidation contribute to skeletal muscle insulin resistance. Cell Metab. 2008 Jan;7(1):45-56. doi: 10.1016/j.cmet.2007.10.013. PMID 18177724
- [Background] Salehzadeh F, Rune A, Osler M, Al-Khalili L. Testosterone or 17beta-estradiol exposure reveals sex-specific effects on glucose and lipid metabolism in human myotubes. J Endocrinol. 2011 Aug;210(2):219-29. doi: 10.1530/JOE-10-0497. Epub 2011 Jun 1. PMID 21632903
- [Background] Hamadeh MJ, Devries MC, Tarnopolsky MA. Estrogen supplementation reduces whole body leucine and carbohydrate oxidation and increases lipid oxidation in men during endurance exercise. J Clin Endocrinol Metab. 2005 Jun;90(6):3592-9. doi: 10.1210/jc.2004-1743. Epub 2005 Mar 8. PMID 15755861
- [Background] Krssak M, Falk Petersen K, Dresner A, DiPietro L, Vogel SM, Rothman DL, Roden M, Shulman GI. Intramyocellular lipid concentrations are correlated with insulin sensitivity in humans: a 1H NMR spectroscopy study. Diabetologia. 1999 Jan;42(1):113-6. doi: 10.1007/s001250051123. PMID 10027589
- [Background] Franklin RM, Kanaley JA. Intramyocellular lipids: effect of age, obesity, and exercise. Phys Sportsmed. 2009 Apr;37(1):20-6. doi: 10.3810/psm.2009.04.1679. PMID 20048484
- [Background] Goodpaster BH, Kelley DE, Wing RR, Meier A, Thaete FL. Effects of weight loss on regional fat distribution and insulin sensitivity in obesity. Diabetes. 1999 Apr;48(4):839-47. doi: 10.2337/diabetes.48.4.839. PMID 10102702
- [Background] Lara-Castro C, Newcomer BR, Rowell J, Wallace P, Shaughnessy SM, Munoz AJ, Shiflett AM, Rigsby DY, Lawrence JC, Bohning DE, Buchthal S, Garvey WT. Effects of short-term very low-calorie diet on intramyocellular lipid and insulin sensitivity in nondiabetic and type 2 diabetic subjects. Metabolism. 2008 Jan;57(1):1-8. doi: 10.1016/j.metabol.2007.05.008. PMID 18078853
- [Background] Tamura Y, Tanaka Y, Sato F, Choi JB, Watada H, Niwa M, Kinoshita J, Ooka A, Kumashiro N, Igarashi Y, Kyogoku S, Maehara T, Kawasumi M, Hirose T, Kawamori R. Effects of diet and exercise on muscle and liver intracellular lipid contents and insulin sensitivity in type 2 diabetic patients. J Clin Endocrinol Metab. 2005 Jun;90(6):3191-6. doi: 10.1210/jc.2004-1959. Epub 2005 Mar 15. PMID 15769987
- [Background] Mahmood S, Taketa K, Imai K, Kajihara Y, Imai S, Yokobayashi T, Yamamoto S, Sato M, Omori H, Manabe K. Association of fatty liver with increased ratio of visceral to subcutaneous adipose tissue in obese men. Acta Med Okayama. 1998 Aug;52(4):225-31. doi: 10.18926/AMO/31297. PMID 9781273
- [Background] Lewis MC, Phillips ML, Slavotinek JP, Kow L, Thompson CH, Toouli J. Change in liver size and fat content after treatment with Optifast very low calorie diet. Obes Surg. 2006 Jun;16(6):697-701. doi: 10.1381/096089206777346682. PMID 16756727
- [Background] Hall KD. Predicting metabolic adaptation, body weight change, and energy intake in humans. Am J Physiol Endocrinol Metab. 2010 Mar;298(3):E449-66. doi: 10.1152/ajpendo.00559.2009. Epub 2009 Nov 24. PMID 19934407
- [Background] Wells GD, Noseworthy MD, Hamilton J, Tarnopolski M, Tein I. Skeletal muscle metabolic dysfunction in obesity and metabolic syndrome. Can J Neurol Sci. 2008 Mar;35(1):31-40. doi: 10.1017/s0317167100007538. PMID 18380275
- [Background] Bergman RN, Ider YZ, Bowden CR, Cobelli C. Quantitative estimation of insulin sensitivity. Am J Physiol. 1979 Jun;236(6):E667-77. doi: 10.1152/ajpendo.1979.236.6.E667. PMID 443421
- [Background] Elia M, Livesey G. Energy expenditure and fuel selection in biological systems: the theory and practice of calculations based on indirect calorimetry and tracer methods. World Rev Nutr Diet. 1992;70:68-131. doi: 10.1159/000421672. No abstract available. PMID 1292242
- [Derived] Whytock KL, Corbin KD, Parsons SA, Pachori A, Bock CP, Jones KP, Smith JS, Yi F, Xie H, Petucci CJ, Gardell SJ, Smith SR. Metabolic adaptation characterizes short-term resistance to weight loss induced by a low-calorie diet in overweight/obese individuals. Am J Clin Nutr. 2021 Jul 1;114(1):267-280. doi: 10.1093/ajcn/nqab027. PMID 33826697
- See also: Translational Research Institute for Metabolism and Diabetes web page for more information on the study — http://www.tri-md.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overweight/obese participant were recruited to the study to participate in a 28 day low calorie diet (LCD). After 28 days, participants were evaluated for whether they met their expected weight loss targets. If participants met their targets they continued the LCD for a further 28 days and are defined as Overweight/Obese With no Drug. If participants did not reach their weight loss target they continued with LCD with an addition of phentermine and are defined as Overweight/Obese With Phentermine
Groups:
- Overweight/Obese With no Drug: After screening, overweight (obese subjects (BMI<27 - ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved.
  Low Calorie Diet (LCD): A Diet History Questionnaire will be completed, and the subjects will have dietary counseling and be provided shakes. LCD period= continuous for 8 weeks.
- Overweight/Obese With Phentermine: After screening, overweight/obese (BMI 27.0-≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved. Individuals not on track to achieve their target weight by four weeks will receive the drug Phentermine to promote weight loss. Then, following eight weeks LCD (or four weeks LCD + four weeks LCD+Phentermine), in the event that they did not achieve the target weight loss, subjects will be given the option to continue with the LCD + Phentermine for up to an additional 12 weeks, under a doctor's supervision.
  Low Calorie Diet (LCD): A Diet History Questionnaire will be completed, and the subjects will have dietary counseling and be provided shakes. LCD period = continuous for 8 weeks.
  Phentermine: Individuals not on track to achieve their target weight by four weeks will receive the drug Phentermine to promote weight loss. Then, following eight weeks LCD.
Period: Overall Study
Arm/Group | Overweight/Obese With no Drug | Overweight/Obese With Phentermine
Started | 19 | 20
Completed | 19 | 18
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ovweight/Obese With no Drug: After screening, overweight (obese subjects (BMI >27 - ≤40.0) subjects (n=35) will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved.
  Low Calorie Diet (LCD): A Diet History Questionnaire will be completed, and the subjects will have dietary counseling and be provided shakes. The low calorie diet will begin, to continue for a period of 8 weeks.
- Overweigh/Obese With Phentermine: After screening, obese subjects (BMI >27- ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved. Individuals not on track to achieve their target weight by four weeks will receive the drug Phentermine to promote weight loss. Then, following eight weeks LCD (or four weeks LCD + four weeks LCD+Phentermine), in the event that they did not achieve the target weight loss, subjects will be given the option to continue with the LCD + Phentermine for up to an additional 12 weeks, under a doctor's supervision.
  Low Calorie Diet (LCD): See prior information.
  Phentermine: See prior information.
  Protection Against Risk: See prior information.
  .
- Total: Total of all reporting groups
Arm/Group | Ovweight/Obese With no Drug | Overweigh/Obese With Phentermine | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 37.3 [25 to 54] | 43.6 [23 to 56] | 42.3 [23 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Amount of Fat Oxidation at 14 Days
Description: Measured with respiratory quotient obtained with indirect calorimetry
  Expected Results
  * Overweight and obese subjects will show a wide variation in fat oxidation in response to the low calorie diet
  * Approximately one-third of study participants will not meet target weight loss by four weeks
  * Following an overnight fast (prior to and during LCD) individuals that fail to meet the target weight loss will be characterized by decreased whole body fat oxidation and increased carbohydrate oxidation (measured by indirect calorimetry)
Time Frame: Days 0, 14
Measure: Mean (Standard Deviation); unit: Fold change of RQ ratio
Groups:
- Overweight/Obese With no Drug: After screening, overweight (obese subjects (BMI >27 - ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved.
  Low Calorie Diet (LCD): A Diet History Questionnaire will be completed, and the subjects will have dietary counseling and be provided shakes. The low calorie diet will begin, to continue for a period of 8 weeks.
- Overweight/ Obese With Phentermine: After screening, obese subjects (BMI >27 - ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved. Individuals not on track to achieve their target weight by four weeks will receive the drug Phentermine to promote weight loss. Then, following eight weeks LCD (or four weeks LCD + four weeks LCD+Phentermine), in the event that they did not achieve the target weight loss, subjects will be given the option to continue with the LCD + Phentermine for up to an additional 12 weeks, under a doctor's supervision.
  Low Calorie Diet (LCD): See prior information.
  Phentermine: See prior information.
  Protection Against Risk: See prior information.
  .
Arm/Group | Overweight/Obese With no Drug | Overweight/ Obese With Phentermine
Number analyzed (Participants) | 19 | 18
Fold change of RQ ratio | 0.91 (0.05) | 0.94 (0.07)

2. Primary Outcome: Fat Oxidation Rates at 1 Week Intervals
Description: Measured with respiratory quotient using indirect calorimetry
  Expected Results
  * Overweight and obese subjects will show a wide variation in fat oxidation in response to the low calorie diet
  * Approximately one-third of study participants will not meet target weight loss by four weeks
  * Following an overnight fast (prior to and during LCD) individuals that fail to meet the target weight loss will be charaterized by decreased whole body fat oxidation and increased carbohydrate oxidation (measured by indirect calorimetry)
Time Frame: Days 0, 7, 14, 28, 49, 56
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Overweight/ Obese With no Drug: After screening, overweight (obese subjects (BMI >27 - ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved.
  Low Calorie Diet (LCD): A Diet History Questionnaire will be completed, and the subjects will have dietary counseling and be provided shakes. The low calorie diet will begin, to continue for a period of 8 weeks.
Arm/Group | Overweight/ Obese With no Drug | Overweight/ Obese With Phentermine
Number analyzed (Participants) | 19 | 18
Ratio
  Day 0 | 0.867 (0.052) | 0.857 (0.059)
  Day 7 | 0.795 (0.041) | 0.787 (0.039)
  Day 14 | 0.791 (0.036) | 0.801 (0.041)
  Day 28 | 0.808 (0.034) | 0.811 (0.069)
  Day 49 | 0.800 (0.048) | 0.784 (0.044)
  Day 56 | 0.798 (0.048) | 0.785 (0.048)

3. Secondary Outcome: Soleus IMCL Content
Description: Measured with magnetic resonance spectroscopy (MRS)
  Expected results
  * 1H-MRS can measure skeletal muscle (intramyocellular lipid) IMCL content with low test-retest variability
  * 1H-MRS can sensitively monitor reductions (or lack thereof) in skeletal muscle IMCL during caloric restriction
  * Reductions in IMCL will be higher in subjects with lower fasting respiratory quotients (RQ) at baseline/during LCD
Time Frame: Days -7, -1, 14, 56
Measure: Mean (Standard Deviation); unit: ratio of peak height of IMCL to water
Arm/Group | Overweight/ Obese With no Drug | Overweight/ Obese With Phentermine
Number analyzed (Participants) | 19 | 18
ratio of peak height of IMCL to water
  Day -7 | 0.025 (0.010) | 0.032 (0.015)
  Day 0 | 0.028 (0.014) | 0.034 (0.019)
  Day 14 | 0.030 (0.011) | 0.034 (0.011)
  Day 56 | 0.027 (0.014) | 0.034 (0.013)

ADVERSE EVENTS:
Groups:
- Overwight/Obese With Phentermine: After screening, obese subjects (BMI >27 - ≤40.0) subjects will be started on a low calorie diet (approximately 900-1000 kcal/d) until a target weight loss is achieved. Individuals not on track to achieve their target weight by four weeks will receive the drug Phentermine to promote weight loss. Then, following eight weeks LCD (or four weeks LCD + four weeks LCD+Phentermine), in the event that they did not achieve the target weight loss, subjects will be given the option to continue with the LCD + Phentermine for up to an additional 12 weeks, under a doctor's supervision.
  Low Calorie Diet (LCD)
  Phentermine
Arm/Group | Overweight/Obese With no Drug | Overwight/Obese With Phentermine
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes